CLINICAL TRIAL: NCT05015504
Title: Application of Time Restriction Feeding in Patients With Type 2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Collaborators: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1770741-4
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: intermittent fasting; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Single group self comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time restricted feeding (Experimental): The study will consist of three phases. In phase I all study subjects will be in the ad libitum feeding phase for one week followed by Phase II. In Phase II the subjects will be placed on time-restricted fasting (feeding between 4 AM - 4 PM, fasting in the rest of the day) for one week. For phase III (final week), patients will be returned to an ad libitum feeding. The first and third phases will serve as control phases, and the second phase will be the experimental phase
  Interventions: Behavioral: Time restricted feeding

INTERVENTIONS:
Behavioral: Time restricted feeding — In Phase II the study subjects will be placed on time-restricted fasting (feeding between 4 AM - 4 PM, fasting in the rest of the day) for one week.
  Other Names: Ad libitum feeding

SUMMARY:
In this 3-week interventional study, the investigators hypothesize that therapeutic Time-Restricted Feeding in patients with poorly controlled Type 2 diabetes mellitus (T2DM) can improve their mean glucose or estimated glycated hemoglobin levels with the same dose, or even reduced dose, of antidiabetics.

DETAILED DESCRIPTION:
Time-restricted feeding (TRF) has recently gained popularity as a means of reducing body weight and improving glycemia. A recent clinical trial in men who had prediabetes showed that TRF for five weeks significantly reduced fasting insulin concentration and improved the derived oral glucose tolerance test ( OGTT) indexes of beta-cell responsiveness and insulin resistance. However, the effects of TRF have not been studied in patients with poorly controlled Type 2 diabetes mellitus (T2DM). In this 3-week interventional self-controlled clinical trial, the investigators hypothesize that TRF in patients with poorly-controlled T2DM can improve their mean glucose with the same dose/reduced dose of antidiabetics. Potential study subjects will be identified from Endocrinology clinic patients with a diagnosis of poorly controlled type 2 DM (A1c >= 8.0 in the 3 months before enrollment) based on inclusion and exclusion criteria. All study subjects will be in the ad libitum feeding phase for one week, and then will be placed on time-restricted fasting (feeding between 4 AM - 4 PM, fasting in the rest of the day) for the second week. For the third and final week, patients will be returned to the ad libitum feeding phase. The first and third weeks will serve as the control phases, and the second week will be the experimental phase. The mean glucose, serum triglyceride levels, insulin resistance, and body weights will be compared between the two phases. Results of this clinical study may demonstrate a low-cost and practical way of diabetic control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 65 years
* With the diagnosis of type 2 diabetes
* A1c >= 8.0 on the most recent test in the 3 months before enrollment
* Have been on stable antidiabetics in the 3 months before enrollment
* OhioHealth Patient

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Severe hypoglycemic episodes (defined as having low blood glucose levels that requires assistance from another person to treat) in the past 12 months
* Unable to give informed consent
* Currently enrolled in another therapeutic study
* Thyroid dysfunction, as defined by abnormal thyroid function test results within the past 6 months
* Advanced stage of renal (stage 4 or above) or hepatic (cirrhosis) or respiratory (needs oxygen) or heart failure (NYHA class 3 or above)
* Active infection or malignancy
* Dementia, or other significant mental impairment that would, in the opinion of the investigator, impede patient self-reporting
* Clinician-reported history of patient non-adherence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
mean glucose | in one week of time restricted feeding
  change in mean glucose
estimated hemoglobin A1c levels | in one week of time restricted feeding
  change in estimated hemoglobin A1c levels

SECONDARY OUTCOMES:
Insulin resistance | in one week of time restricted feeding
  change in Insulin resistance is represented by the homeostatic model of assessment of insulin resistance
serum triglyceride levels | in one week of time restricted feeding
  change serum triglycerides are measured by a fasting lipid panel
body weight | in one week of time restricted feeding
  change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjie Mao, MD, PhD, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth Castrop Health Center, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zubrzycki A, Cierpka-Kmiec K, Kmiec Z, Wronska A. The role of low-calorie diets and intermittent fasting in the treatment of obesity and type-2 diabetes. J Physiol Pharmacol. 2018 Oct;69(5). doi: 10.26402/jpp.2018.5.02. Epub 2019 Jan 21. PMID 30683819
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Barnosky AR, Hoddy KK, Unterman TG, Varady KA. Intermittent fasting vs daily calorie restriction for type 2 diabetes prevention: a review of human findings. Transl Res. 2014 Oct;164(4):302-11. doi: 10.1016/j.trsl.2014.05.013. Epub 2014 Jun 12. PMID 24993615